CLINICAL TRIAL: NCT05454670
Title: The Effect of Collagen Matrix Graft on Postoperative Palatal Fistula Formation After Cleft Palate Repair: A Randomized Controlled Study
Brief Title: Effect of Collagen Matrix Graft on Palatal Fistula Formation After Cleft Palate Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lagos State University (Other)
Collaborators: University of Lagos, Nigeria (Other)
Responsible Party: Principal Investigator, Egbunah Uchenna Patrick, Senior Registrar, University of Lagos, Nigeria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ADM/DST/HREC/VOL.XVII/763
Record Dates: First submitted 2022-07-02; First posted 2022-07-12 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Cleft Lip and Cleft Palate; Cleft Lip, Cleft Alveolus and Cleft Palate; Cleft Palate
Keywords: cleft palate; palatal fistula; collagen graft
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Intervention Model Description: The study will be a parallel randomized controlled study involving two groups of participants. The test group will include participants with who will undergo cleft palate repair with collagen graft used as superpositional graft between the nasal mucosa/muscle layer and the oral mucosa layer when two-flap palatoplasty is performed while the control group will include participants who undergo two-flap palatoplasty without the use of collagen graft
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study will be a double-blind randomized controlled study. After random allocation, the participants (parents/ patients) will be unaware of the study group they belong to. Also, the surgeon assessing postoperative outcomes will not perform the surgery and will be unaware of the study group of the participant being examined. Since the collagen graft will be placed between the nasal/ muscular layers and the oral layer, it is expected that after apposition of the oral layer, no collagen matrix will be visible intraorally to reveal the study group of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The intervention will be primary cleft palate repair using resorbable collagen matrix graft as superpositional graft during approximation of the nasal mucosa and muscular layer in cleft palate repair. The collagen graft with be inserted between the nasal mucosa/ muscular layer and the oral mucosa layer during two-flap palatoplasty.
  Interventions: Procedure: Two-flap palatoplasty
- Control group (Active Comparator): The intervention will be primary cleft palate repair using two-flap palatoplasty technique without collagen graft
  Interventions: Procedure: Two-flap palatoplasty

INTERVENTIONS:
Procedure: Two-flap palatoplasty — Two-flap palatoplasty used to correct cleft palate defect. The cleft palate is closed by separation of the nasal and the oral mucosa layers. Then approximation of the nasal mucosa layer, muscle layer is secured in the posterior palate and then the oral mucosa layer is secured

SUMMARY:
Palatal fistulas are a major burden to surgeons and patients in the management of cleft palate. Their high rate of occurrence and recurrence makes them particularly challenging even to the highly skilled surgeon. Prevention of postoperative palatal fistula is therefore of paramount importance.

Closure of the nasal mucosa under tension has been proposed as a major cause of palatal fistula formation. However, depending on the presentation of the cleft palate, it may be impossible to achieve surgical closure with minimal tension. Till date, there is no universally acceptable method of preventing palatal fistula formation following cleft palate repair. And although the use of pre-surgical appliances such as Latham appliance and the use of local and distant tissues to achieve two layer closure have been proposed, the use of a superpositional collagen graft may also be used to achieve closure of the nasal mucosa with minimal or no tension during cleft palate repair.

Collagen grafts have the added advantage of being more patient friendly compared to the Latham appliance which requires an initial surgery for appliance insertion before surgical cleft palate repair. They are also less technique sensitive compared to the use of local and distant tissues.

The investigators therefore aim to provide high level scientific evidence of the effectiveness of collagen graft in the prevention of postoperative palatal fistula.

ELIGIBILITY:
Inclusion Criteria:

* Non-syndromic cleft palate
* Must be between nine months to two years
* Must have not previously had cleft palate surgery
* Must consent to participate in the study

Exclusion Criteria:

* All blood dyscrasias
* All connective tissue dysfunctions

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative palatal fistula | 24 hours post operatively
  Palatal fistula will be defined as a patency between the oral and nasal cavities developing postoperatively anywhere along the primary or secondary palate
Number of participants with postoperative palatal fistula | Seven days post operatively
  Palatal fistula will be defined as a patency between the oral and nasal cavities developing postoperatively anywhere along the primary or secondary palate
Number of participants with postoperative palatal fistula | Two weeks post operatively
  Palatal fistula will be defined as a patency between the oral and nasal cavities developing postoperatively anywhere along the primary or secondary palate
Number of participants with postoperative palatal fistula | One month post operatively
  Palatal fistula will be defined as a patency between the oral and nasal cavities developing postoperatively anywhere along the primary or secondary palate

SECONDARY OUTCOMES:
Number of participants with wound dehiscence | 24 hours post operatively
  Wound dehiscence will be defined as partial or total separation of previously approximated and sutured surgical wound edges with or without palatal fistula formation.
Number of participants with wound dehiscence | Seven days post operatively
  Wound dehiscence will be defined as partial or total separation of previously approximated and sutured surgical wound edges with or without palatal fistula formation.
Number of participants with wound dehiscence | Two weeks post operatively
  Wound dehiscence will be defined as partial or total separation of previously approximated and sutured surgical wound edges with or without palatal fistula formation.
Number of participants with wound dehiscence | One month post operatively
  Wound dehiscence will be defined as partial or total separation of previously approximated and sutured surgical wound edges with or without palatal fistula formation.
Number of participants with surgical site inflammation | 24 hours post operatively
  Surgical site inflammation will be defined as tenderness, redness, swelling and/or differential warmth from surgical site.
Number of participants with surgical site inflammation | Seven days post operatively
  Surgical site inflammation will be defined as tenderness, redness, swelling and/or differential warmth from surgical site.
Number of participants with surgical site inflammation | Two weeks post operatively
  Surgical site inflammation will be defined as tenderness, redness, swelling and/or differential warmth from surgical site.
Number of participants with surgical site inflammation | One month post operatively
  Surgical site inflammation will be defined as tenderness, redness, swelling and/or differential warmth from surgical site.
Number of participants with surgical site infection | 24 hours post operatively
  Surgical site infection will be defined as tenderness and purulent discharge and/or foul smelling odor from surgical site
Number of participants with surgical site infection | Seven days post operatively
  Surgical site infection will be defined as tenderness and purulent discharge and/or foul smelling odor from surgical site
Number of participants with surgical site infection | Two weeks post operatively
  Surgical site infection will be defined as tenderness and purulent discharge and/or foul smelling odor from surgical site
Number of participants with surgical site infection | One month post operatively
  Surgical site infection will be defined as tenderness and purulent discharge and/or foul smelling odor from surgical site
Surgeon satisfaction | within the first 24 hours post operatively
  Surgeon satisfaction will assess surgeons' opinion on surgery time (normal/ extended), difficulty of procedure (not difficult/ increased difficulty) and inadvertent tearing of the nasal mucosa (absent/ present).

CONTACTS AND LOCATIONS:
Locations (1):
- Lagos University Teaching Hospital, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided